CLINICAL TRIAL: NCT04466033
Title: Evaluation of the Safety and Performance of Magneto Microcatheter for Endovascular Thrombectomy in Patients With Acute Ischemic Stroke
Brief Title: Evaluation of the Safety and Performance of Magneto Microcatheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Magneto Thrombectomy Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14-CLN002
Record Dates: First submitted 2020-07-05; First posted 2020-07-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magneto Microcatheter (Experimental)
  Interventions: Device: Magneto Microcatheter

INTERVENTIONS:
Device: Magneto Microcatheter — All patients will be treated with Magneto Microcatheter

SUMMARY:
A prospective, open label single arm feasibility study to evaluate the safety and performance of the Magneto Microcatheter in patients diagnosed with acute ischemic stroke and planned for thrombectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs consistent with acute ischemic stroke
2. Patient with Acute Ischemic Stroke within 24 hours from symptoms o
3. Age 18-85 years old
4. Consent process is completed per international and local regulations

Exclusion Criteria:

1. Known use of cocaine or other vasoactive substance
2. Known bleeding diathesis
3. Any known hemorrhagic or coagulation deficiency.
4. Current use of oral anticoagulants with International Normalized Ratio (INR) > 3;
5. PTT (Partial Thromboplastin Time)>2 at screening
6. Uncontrolled hypertension (Systolic blood pressure>185 or Diastolic blood pressure>110) refractory to pharmacological management
7. Pregnant or lactating female
8. CT scan or MRI with evidence of acute intracranial hemorrhage, ASPECT score<6, mass effect and/or intracranial tumor
9. Angiographic evidence of either carotid dissection or vasculitis at the target site or any condition that may limit device access to the target site (i.e high grade stenosis) per the treating physician's discretion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety of Magneto Microcatheter in the acute post procedure duration by assessing the incidence of device related Serious Adverse Events within 24 hours post procedure | 24 hours
  Occurrence of device related Serious Adverse Events

SECONDARY OUTCOMES:
Evaluation of the safety of Magneto Microcatheter by assessing the incidence of device related Serious Adverse Events within 90 days post procedure | 90 days
  Occurrence of device related Serious Adverse Events
Evaluation of the performance of Magneto Microcatheter by assessing its ability to remove the clot and evaluating its ease of use | During Procedure
  Assessment of device performance in clot removal (TICI scale to evaluate revascularization) and ease of use (questionnaire that will be completed by the treating physician post procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Marzelik, Principal Investigator — Sheba Medical Center; Dr.Amsalem, Principal Investigator — Shaare Zedek, Israel
Locations (3):
- National Institute of Mental Health, Neurology and Neurosurgery), Budapest, Hungary
- Israel (2):
  - Shaare Zedek, Jerusalem
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No